CLINICAL TRIAL: NCT00151411
Title: The Effect of Combination Therapy With Lifestyle Intervention and Metformin in Females With Polycystic Ovary Syndrome
Brief Title: Lifestyle Intervention and Metformin for Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2003-172; HD-02-012
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome (PCOS); Anovulation; Elevated Testosterone
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin
  Interventions: Drug: Metformin; Behavioral: Lifestyle Intervention
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Metformin — Medication was initiated in a step-up fashion every five days, from one tablet per day to four (500 mg per tablet).
  Arms: Metformin
Drug: Placebo — Placebo
  Arms: Placebo
Behavioral: Lifestyle Intervention — A combined intervention of diet and exercise was employed with the goal of achieving an average weight loss of at least 7% of initial body weight over six months with a prescription of 150 min/week of exercise combined with a low-calorie diet.

SUMMARY:
The purpose of this study is to determine if the combination therapy of lifestyle intervention and use of Metformin together will improve ovulation induction and hyperandrogenemia in women with polycystic ovary syndrome, by gathering data from adult and adolescent females.

DETAILED DESCRIPTION:
PCOS is characterized by excess circulating androgen levels and chronic anovulation. PCOS is also characterized by insulin resistance and hyperinsulinemia. Several recent studies in a variety of non-hospital based populations have provided evidence that the incidence of hyperandrogenic chronic anovulation is in the range of 4-6% of the female population. Improvements in insulin sensitivity in women with PCOS, either through lifestyle changes or through pharmaceutical intervention, have consistently resulted in a marked improvement in the reproductive and metabolic abnormalities in PCOS. The primary objective in the adult female population is to determine that combination therapy will improve ovulatory frequency. Secondary objective is to improve circulating hyperandrogenemia and insulin sensitivity then single agent therapy. The primary objective of the adolescent population is to determine that the combination therapy will improve hyperandrogenemia. Secondary objective is to improve ovulatory frequency and insulin sensitivity than just the use of a single agent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intermenstrual periods of greater than or equal to 45 days or a total of 8 or less periods per year
* Elevated testosterone levels
* General good health
* Off of current medications which may confound response to study medications

Exclusion Criteria:

* Pregnancy
* Lactose Intolerance
* Medical Contraindications
* Elevated Prolactin, 17hydroxyprogesterone, or Follicle stimulating hormone blood tests
* Diabetes, liver, heart, kidney or uncorrected thyroid disease

Ages: 12 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Ladson G, Dodson WC, Sweet SD, Archibong AE, Kunselman AR, Demers LM, Lee PA, Williams NI, Coney P, Legro RS. Effects of metformin in adolescents with polycystic ovary syndrome undertaking lifestyle therapy: a pilot randomized double-blind study. Fertil Steril. 2011 Jun 30;95(8):2595-8.e1-6. doi: 10.1016/j.fertnstert.2011.05.048. PMID 21704212
- [Derived] Ladson G, Dodson WC, Sweet SD, Archibong AE, Kunselman AR, Demers LM, Williams NI, Coney P, Legro RS. The effects of metformin with lifestyle therapy in polycystic ovary syndrome: a randomized double-blind study. Fertil Steril. 2011 Mar 1;95(3):1059-66.e1-7. doi: 10.1016/j.fertnstert.2010.12.002. Epub 2010 Dec 30. PMID 21193187
- See also: Click here for more information about this study — http://www.pennstatehershey.org/web/obgyn/patientcare/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin 2000mg/d (2 500mg tablets taken twice a day) initiated in a step-up fashion
- Placebo: Placebo (2 tablets twice a day) initiated in a step-up fashion
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 55 | 59
Completed | 22 | 16
Not Completed | 33 | 43
Not completed — Lost to Follow-up | 15 | 19
Not completed — Withdrawal by Subject | 12 | 20
Not completed — Adverse Event | 6 | 0
Not completed — Pregnancy | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 55 | 59 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 59 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4.5) | 28.8 (4.6) | 28.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 59 | 114
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 59 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change in Testosterone After 6 Months of Treatment
Time Frame: baseline and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 55 | 59
ng/dL | -2.1 [-12.1 to 7.9] | -6.4 [-16.9 to 4.1]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.54, Mixed Models Analysis; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-9.9 to 18.4]

2. Secondary Outcome: Ovulation Rate
Description: Count of ovulations per subject during the treatment period.
Time Frame: 6 months
Population: A total of 76 patients with daily urine collections.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 37 | 39
Participants
  0 ovulations | 10 | 19
  1 ovulation | 6 | 5
  2 ovulations | 4 | 7
  3 ovulations | 7 | 3
  4 ovulations | 4 | 2
  5 ovulations | 1 | 0
  6+ ovulations | 5 | 3
Statistical Analysis 1: Comparison: Metformin vs Placebo; This statistical analysis models the probability of ovulation; Test type: Superiority; p = 0.07, Zero-altered negative binomial model; Rate Ratio = 2.5, 95% CI 2-sided [0.9 to 6.6] — Placebo is the reference group, i.e. for the rate ratio, Metformin represents the numerator and Placebo the denominator
Statistical Analysis 2: Comparison: Metformin vs Placebo; This statistical analysis models the count of ovulations provided a woman actually ovulated; Test type: Superiority; p = 0.51, Zero-altered negative binomial model; rate ratio = 1.2, 95% CI 2-sided [0.7 to 1.9] — Placebo is the reference group, i.e. for the rate ratio, Metformin represents the numerator and Placebo the denominator

3. Secondary Outcome: Change in Insulin Sensitivity Index After 6 Months of Treatment
Time Frame: baseline and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 55 | 59
index | 1.9 [-1.0 to 4.8] | -2.7 [-6.2 to 0.9]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [0.1 to 9.0]

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/59
Other Adverse Events (participants affected / at risk) | 38/55 | 33/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=55) | Placebo (N=59)
Diarrhea (Gastrointestinal disorders) | 19 (78) | 6 (22)
stomach/abdominal pain or discomfort (Gastrointestinal disorders) | 6 (9) | 7 (16)
nausea and/or vomiting (Gastrointestinal disorders) | 9 (27) | 7 (18)
flatulence (Gastrointestinal disorders) | 2 (5) | 3 (3)
flu (Gastrointestinal disorders) | 8 (12) | 4 (4)
common cold/respiratory tract infection (Infections and infestations) | 12 (23) | 13 (19)
dizziness (Nervous system disorders) | 3 (5) | 3 (3)
headache/migraine (Nervous system disorders) | 12 (42) | 11 (16)
fatigue (Nervous system disorders) | 2 (2) | 4 (4)
altered mood/mood swings (Nervous system disorders) | 0 (0) | 5 (6)
dysmenorrhea/cramps (Reproductive system and breast disorders) | 7 (14) | 9 (19)
vaginal infection (Reproductive system and breast disorders) | 3 (3) | 3 (3)
bladder infection (Renal and urinary disorders) | 1 (2) | 3 (9)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (7) | 9 (17)
hair loss (General disorders) | 3 (3) | 0 (0)
allergic reaction (General disorders) | 0 (0) | 3 (3)
dental issues (General disorders) | 3 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No